CLINICAL TRIAL: NCT02785419
Title: Targeted Engagement of the Motor Action Selection Network During Arm Rehabilitation After Stroke
Brief Title: Action Selection and Arm Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Jill Stewart, PT, PhD, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032516
Record Dates: First submitted 2016-05-09; First posted 2016-05-27 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Rehabilitation; Upper Extremity; Physical Therapy
MeSH Terms: conditions — Stroke

ARMS (1):
- Arm Training with Action Selection (Experimental): Task-oriented, functional arm training with the addition of action selection cues to practice. All participants receive the same arm training intervention.
  Interventions: Behavioral: Arm Training with Action Selection

INTERVENTIONS:
Behavioral: Arm Training with Action Selection — Treatment occurs in 1.5 hour sessions, 5 times a week for 3 weeks. In each treatment session, you will practice functional tasks with your weaker arm and hand. Additionally, you will be given cues on a computer screen that dictate your movement response (action selection). Practice will be scaled to match your current level of function and progressed over time as able.
  Other Names: Functional task practice; Arm rehabilitation

SUMMARY:
After stroke, individuals often have persistent difficulty using the arm and hand in everyday functional tasks that reduces quality of life. Currently available rehabilitation techniques are not adequate and new protocols are needed that are based on an understanding of how brain regions work together to produce skilled movement. This research project aims to improve our understanding of how the brain controls movement after stroke and determine whether a period of motor practice that targets specific brain regions through the addition of action selection demands leads to improved arm function. We hypothesize that arm motor function and the ability to efficiently activate the action selection motor circuit during movement will improve after training.

DETAILED DESCRIPTION:
Rehabilitation of arm impairment after stroke includes the repetitive practice of functional tasks. In healthy adults, planning plays a vital role in the control of skilled movement, however, the behavioral and neural correlates of planning have largely been unexplored in individuals recovering from stroke. Action selection is an important motor planning process that engages dorsal premotor cortex (PMd) in controls. While PMd activation is a commonly reported neural correlate of motor recovery after stroke, the role of PMd in action selection and motor training are not known. Therefore, the purpose of this study is to determine the effect of training that includes action selection demands on the behavioral and neural correlates of movement after stroke. Thirty-eight individuals in the chronic phase of stroke will be recruited. After completion of clinical measures of impairment and function, all participants with stroke will complete a motor action selection task and functional MRI followed by arm training. Arm training will consist of three weeks (15 sessions) of arm motor training (1.5 hours per session) that includes action selection demands on movement. Follow-up clinical testing will occur at the end of treatment and three weeks later.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Had stroke at least 6 months ago
* Right-hand dominant prior to stroke
* Some continued arm and hand weakness
* Some ability to move the arm and hand that is weaker from the stroke

Exclusion Criteria:

* Acute medical issues that would interfere with participation
* Another neurologic diagnosis that may impact movement (e.g. Parkinson's Disease)
* Cannot undergo MRI scanning
* Severe apraxia or hemispatial neglect
* Pain in the arm that interferes with movement
* Difficulty maintaining attention or following directions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | Change from baseline to end of treatment (3 weeks)
  Behavioral assessment of arm function. Scores range from 0 to 57 with a higher score equating to better function.
Brain activation during functional MRI | Change from baseline to end of treatment (3 weeks)
  Brain activation during movement will be captured with functional MRI. Analyses will investigate changes in magnitude of activation.
Brain connectivity during functional MRI | Change from baseline to end of treatment (3 weeks)
  Brain activation during movement will be captured with functional MRI. Analyses will investigate changes in connectivity between brain regions.

SECONDARY OUTCOMES:
Upper Extremity Fugl-Meyer Motor Assessment | Change from baseline to end of treatment (3 weeks)
Stroke Impact Scale Hand Domain | Change from baseline to end of treatment (3 weeks)
Box & Blocks Test | Change from baseline to end of treatment (3 weeks)
9-Hole Peg Test | Change from baseline to end of treatment (3 weeks)
Grip Strength | Change from baseline to end of treatment (3 weeks)
Confidence in Arm and Hand Movements Questionnaire | Change from baseline to end of treatment (3 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States